CLINICAL TRIAL: NCT05617664
Title: Is Mirabegron 25 mg Safe and Effective in Treatment of Primary Nocturnal Enuresis as Regard Oral Desmopressin 120 mcg?
Brief Title: Mirabegron 25 mg for Treatment of Primary Nocturnal Enuresis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Hosam Abu El-nasr, lecturer of urology, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: treatment of primary nocturnal
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Nocturnal Enuresis
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Deamino Arginine Vasopressin; mirabegron; Tablets; Behavior Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients with primary nocturnal enuresis will be followed up with behavioral therapy alone. (Placebo Comparator)
  Interventions: Behavioral: behavioral therapy alone
- patients with primary nocturnal enuresis will take desmopressin 120 mcg oral tablets. (Active Comparator)
  Interventions: Drug: desmopressin 120 mcg oral tablets
- patients with PNE will take mirabegron 25 mg oral tablets. (Active Comparator)
  Interventions: Drug: Mirabegron 25 MG Oral Tablet, Extended Release

INTERVENTIONS:
Drug: desmopressin 120 mcg oral tablets — treatment for three months then will stop
  Arms: patients with primary nocturnal enuresis will take desmopressin 120 mcg oral tablets.
Drug: Mirabegron 25 MG Oral Tablet, Extended Release — treatment for three months then will stop
  Arms: patients with PNE will take mirabegron 25 mg oral tablets.
Behavioral: behavioral therapy alone — no medications will be given to the patient
  Arms: patients with primary nocturnal enuresis will be followed up with behavioral therapy alone.

SUMMARY:
Investigators will study the efficacy and safety of mirabegron25 in treatment of primary nocturnal enuresis in comparison to oral desmopressin 120 mcg and behavioral therapy

DETAILED DESCRIPTION:
No doubt that nocturnal enuresis is one of the commonest types of urinary incontinence which affect children and always run in family . Nocturnal enuresis occurs at the age of 5 years with leakage of urine involuntarily during sleep for two times or more per week in three consecutive months not due to congenital or acquired cause. Nocturnal enuresis can be categorized into primary or secondary depending on occurrence of bed dryness for more than six months or not .

Nocturnal enuresis affects 15% to 20 % of children at five years old mainly due to delay of bladder development and function more in male children with presence of family history in half of cases but 15% of children with enuresis recover spontaneously every year .

limitation of fluid intake, urotherapy and bedwetting alarms are non-pharmacological treatments of nocturnal enuresis while the mostly used drugs for treatment of NE are tricyclic antidepressants(Imipramine®) an arginine vasopressin analog (Desmopressin®) and anticholinergic drugs . Enuresis alarms have pitfalls which disgust a lot of patients as skin irritation, sleep disturbances of other family members and failure to wake the child so that about 30% of patients stop its usage .

Desmopressin is approved as a first-line drug therapy for nocturnal enuresis , but a lot of series declared that monotherapy with desmopressin has little efficacy in treating patients which have bladder storage dysfunction furthermore, high recurrence rate after treatment cessation .

The International Children's Continence Society (ICCS) recommended combination therapy for treatment of primary nocturnal enuresis after failure of first line therapy with desmopressin or enuresis alarms . As regard anticholinergic drugs, oxybutynin was firstly prescribed then tolterodine with less side effects and lately solifenacin . Cognitive impairment as a neurological side effect was authenticated for oxybutynin and other side effects (e.g. headache, dry mouth, behavior change, flushed cheeks, constipation, and blurred vision) were unbearable to many children and impulsed them to stop treatment early .

Mirabegron, a b3-adrenoceptor (b3-AR) agonist was the answer to the question about a drug that can relax detrusor muscle and increasing bladder capacity without the limitations of anti-cholinergic drugs. Mirabegron is the first b3-AR agonist to be prescribed clinically for OAB symptoms in adults and showed promising outcomes . while it is not licensed to be used in children with overactive bladder, some early reports declared its efficacy and tolerability in children .

So investigators will study the efficacy and safety of mirabegron in treatment of primary nocturnal enuresis

ELIGIBILITY:
Inclusion Criteria:

* primary nocturnal enuresis,
* negligible daytime wetting,
* wet at least 4 times over 4 weeks
* normal clinical examination with no neurological or urological cause for the enuresis

Exclusion Criteria:

* secondary enuresis, polysymptomatic
* neurologic bladder, neurological disorders,
* urinary incontinence disorders
* previous anti NE drugs.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
nocturnal enuresis improvement rate | four months
  decrease number of nights or absent nights the patient get wet

SECONDARY OUTCOMES:
side effects of drugs used | three months
  appearance of any side effect of desmopressin or mirabegron

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospitals, Banhā, Qaliopia, Egypt

REFERENCES:
- [Result] Bayne AP, Skoog SJ. Nocturnal enuresis: an approach to assessment and treatment. Pediatr Rev. 2014 Aug;35(8):327-34; quiz 335. doi: 10.1542/pir.35-8-327. PMID 25086164
- [Result] Nitti VW, Rosenberg S, Mitcheson DH, He W, Fakhoury A, Martin NE. Urodynamics and safety of the beta(3)-adrenoceptor agonist mirabegron in males with lower urinary tract symptoms and bladder outlet obstruction. J Urol. 2013 Oct;190(4):1320-7. doi: 10.1016/j.juro.2013.05.062. Epub 2013 May 30. PMID 23727415
- [Result] Herschorn S, Barkin J, Castro-Diaz D, Frankel JM, Espuna-Pons M, Gousse AE, Stolzel M, Martin N, Gunther A, Van Kerrebroeck P. A phase III, randomized, double-blind, parallel-group, placebo-controlled, multicentre study to assess the efficacy and safety of the beta(3) adrenoceptor agonist, mirabegron, in patients with symptoms of overactive bladder. Urology. 2013 Aug;82(2):313-20. doi: 10.1016/j.urology.2013.02.077. Epub 2013 Jun 13. PMID 23769122
- [Result] Blais AS, Nadeau G, Moore K, Genois L, Bolduc S. Prospective Pilot Study of Mirabegron in Pediatric Patients with Overactive Bladder. Eur Urol. 2016 Jul;70(1):9-13. doi: 10.1016/j.eururo.2016.02.007. Epub 2016 Feb 11. PMID 26876327
- [Result] Park JS, Lee YS, Lee CN, Kim SH, Kim SW, Han SW. Efficacy and safety of mirabegron, a beta3-adrenoceptor agonist, for treating neurogenic bladder in pediatric patients with spina bifida: a retrospective pilot study. World J Urol. 2019 Aug;37(8):1665-1670. doi: 10.1007/s00345-018-2576-0. Epub 2018 Dec 3. PMID 30511212
- [Result] Vande Walle J, Rittig S, Bauer S, Eggert P, Marschall-Kehrel D, Tekgul S; American Academy of Pediatrics; European Society for Paediatric Urology; European Society for Paediatric Nephrology; International Children's Continence Society. Practical consensus guidelines for the management of enuresis. Eur J Pediatr. 2012 Jun;171(6):971-83. doi: 10.1007/s00431-012-1687-7. Epub 2012 Feb 24. PMID 22362256
- [Result] Neveus T, Fonseca E, Franco I, Kawauchi A, Kovacevic L, Nieuwhof-Leppink A, Raes A, Tekgul S, Yang SS, Rittig S. Management and treatment of nocturnal enuresis-an updated standardization document from the International Children's Continence Society. J Pediatr Urol. 2020 Feb;16(1):10-19. doi: 10.1016/j.jpurol.2019.12.020. Epub 2020 Jan 30. PMID 32278657